CLINICAL TRIAL: NCT05129462
Title: Consistency of Immunohistochemical Detecting Assays Using E1L3N and 22C3 Monoclonal Antibodies for Detection of PD-L1 Expression in NSCLC Patients: A Prospective CONFIDENCE Study
Brief Title: Consistency of PD-L1 Detecting Method Between E1L3N and 22C3 Monoclonal Antibodies in NSCLC Patients
Acronym: CONFIDENCE
Status: Completed | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Other Study IDs: CONFIDENCE
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — tissue sample and plasma DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluated the correlation between the qualitative test results of Xiamen Aide PD-L1 antibody reagent (immunohistochemistry) and the efficacy of Keytruda single-agent therapy, and the research data is used to support the registration and marketing of the assessment reagent

ELIGIBILITY:
Inclusion Criteria:

1. ≥18，advanced non-small cell lung cancer confirmed by histopathology, and have received K-drug mono-therapy in the past, the return visit information is complete, with traceable information such as tumor imaging examinations before and after treatment, and the curative effect can be judged;
2. Able to provide FFPE samples with a storage life of 4 years: 6 slices of continuous slices with a thickness of 3-5μm

Exclusion Criteria:

1. Pathological evaluation of the tissue sample has too few tumor cells (total number of tumor cells <100);
2. K-drug mono-therapy is neoadjuvant therapy or adjuvant therapy;
3. Other situations that the investigator thinks are not suitable for participating in this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer who have previously received single-agent K therapy
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-08-05 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Consistency | August 2018- September 2021
  the consistency of PD-L1 expression between monoclonal antibodies of E1L3N and 22C3

SECONDARY OUTCOMES:
PFS | August 2018- September 2021
  Progression free survival time
ORR | August 2018- September 2021
  Objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China